CLINICAL TRIAL: NCT02687672
Title: Transplantation of Purified Autologous Bone Marrow- or Leukapheresis-Derived CD34+ and CD133+ for Patients With Spinal Cord Injuries: A Long-Term Comparative Evaluation of Safety and Efficacy Study.
Brief Title: Transplantation of Autologous Bone Marrow or Leukapheresis-Derived Stem Cells for Treatment of Spinal Cord Injury
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stem Cells Arabia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCA-SCI1
Record Dates: First submitted 2016-02-16; First posted 2016-02-22 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stem Cell Transplantation (Experimental): Injection of leukapheresis-derived, purified, autologous CD34+and CD133+ stem cells
  Interventions: Biological: Stem Cell Transplantation
- Stem Cells (Experimental): Injection of bone marrow-derived, purified, autologous CD34+and CD133+ stem cells.
  Interventions: Biological: Stem Cell Transplantation

INTERVENTIONS:
Biological: Stem Cell Transplantation — Transplantation of autologous stem cells

SUMMARY:
This is a double-armed, Phase I/II trial aims to compare bone marrow and leukapheresis as sources for purified, autologous CD34+ and CD133+ stem cells (SCs), to be utilized in treatment of patients with chronic complete spinal cord injuries (SCI). The study focuses on the safety and efficacy of transplanting un-manipulated, autologous, purified stem cells into the injured spinal cords of patients.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) leads to apoptosis of oligodendrocytes at the injury site resulting in demyelination and neuronal degeneration. This degeneration causes severe functional sensory and motor mutilations that remain an immense challenge to physicians and in which stem cell (SC) transplantation represents a viable alternative. This study is a phase I/II trial aimed at describing a method for treating patients with chronic complete spinal cord injuries (SCI) by utilizing autologous, purified CD34+ and CD133+ stem cells (SCs). The study focuses on the safety and efficacy of transplanting un-manipulated, autologous, purified stem cells in treated patients during a 5-year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from chronic spinal cord injury
* Age of injury ranging from 6-60 months prior to enrollment in this study.
* Ability and willingness to regularly visit Jordan Orthopedic and Spinal Center for post operation follow up.
* Traumatic Injury of spinal cord with complete or partial damage confirmed by MRI.

Exclusion Criteria:

* Injuries less than 6 months old or more than 60 months old
* Non-traumatic injuries (SCI due to inflammation, autoimmune diseases)
* Patients less than 5 or older than 50 years
* Patients suffering from other conditions, including chronic neurological diseases, diabetes mellitus, cardiac/kidney/liver disorders, previous strokes, and previous surgeries unrelated to spinal cord injury.

Ages: 5 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-01; Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Overall clinical improvement in sensory and motor functions using ASIA (American Spinal Cord Injury Association) | 60 months

SECONDARY OUTCOMES:
Improvement in urine and stool incontinence using a questionnaire | 6 months
Functional improvement in impotence and previous sexual erection status (male patients) using a questionnaire | 6 months
Improvement in quality of life using a questionnaire | 6 months
Improvement in personal independence and productivity using questionnaire | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Stem Cells Arabia, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided